CLINICAL TRIAL: NCT06960785
Title: Evaluation of Refractive Outcomes in Patients Undergoing PRESBYOND Using the MEL90 Excimer Laser
Status: Not yet recruiting | Type: Observational
Sponsor: Carl Zeiss Meditec AG (Industry)
Collaborators: GCP-Service International Ltd. & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: GPAS-REF-024-02
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PRESBYOND: Participants in this group will receive a personalized laser eye surgery for the correction of presbyopia (Presbyond). The treatment is planned individually for each patient and performed on both eyes. It involves creating a corneal flap with a femtosecond laser, followed by reshaping the cornea with an excimer laser to improve vision at different distances. One eye is mainly corrected for distance and the other for near vision, allowing the brain to combine both images and support everyday visual tasks without glasses.
  Interventions: Device: MEL90 excimer laser - PRESBYOND

INTERVENTIONS:
Device: MEL90 excimer laser - PRESBYOND — Participants will undergo laser eye surgery in both eyes using the PRESBYOND method. First, a thin flap is created on the surface of the eye using a femtosecond laser. Then, a second laser (excimer laser) reshapes the cornea to improve vision at near, intermediate, and far distances.
  The treatment is similar to monovision techniques, where one eye is mainly corrected for distance and the other for near vision. However, PRESBYOND differs by adjusting the depth of focus in each eye individually, allowing the brain to better combine the two images in the intermediate range-this area is called the "Blend Zone." This approach helps preserve natural binocular (3D) vision, contrast sensitivity, and depth perception. Most patients adapt well and quickly to this type of correction. The procedure is customized based on each patient's age and eye characteristics.

SUMMARY:
The goal of this clinical trial is to collect information on vision outcomes in people aged 45 to 65 who have difficulty seeing clearly at near distances due to aging (a condition called presbyopia). All participants will receive the same treatment: laser eye surgery with the PRESBYOND method using the MEL 90 excimer laser.

The main questions this study aims to answer are:

* How well do patients see at distance, intermediate, and near after treatment?
* How satisfied are patients with their vision after surgery?

Participants will:

* Attend seven visits over six months (before surgery and after surgery at 1 day, 1 week, 1 month, 3 months, and 6 months)
* Undergo laser eye surgery with PRESBYOND
* Complete vision tests and questionnaires about their experience

There is no comparison group in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 45 and 65 years old
2. Scheduled to undergo bilateral LASIK treatment with PRESBYOND
3. Preoperative corrected distance visual acuity of 20/20 Snellen or better in each eye
4. Normal corneal topography in each eye
5. Discontinue use of contact lenses at least 1 month for hard contacts and 1 week for soft lenses prior to the preoperative examination
6. Residual stromal thickness ≥250 microns in each eye
7. Availability, willingness, to comply with examination follow up visits
8. Signed informed consent and data protection documents
9. Patients successfully passed the tolerance test

Exclusion Criteria:

1. Mixed astigmatism in any eye
2. Irregular corneal astigmatism in any eye
3. Clinically significant ocular surface disease in any eye
4. History of ocular surgery, ocular pathology, or other significant ocular findings that, in the Investigator's opinion, may increase the patient's risk for corneal refractive surgery or affect potential visual outcomes in each eye
5. Prior corneal refractive surgery (SMILE, LASIK, LASEK, RK, PRK, etc,) in each eye
6. Amblyopia, strabismus, nystagmus, forme fruste keratoconus in any eye
7. Clinically significant pupil abnormalities in any eye
8. Use of systemic or ocular medications that may affect visual outcomes
9. Systemic pathology that may affect the results of the study
10. Pregnancy or being treated for conditions associated with hormonal fluctuation
11. Participation in another clinical trial in the last 30 days

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants scheduled to undergo laser eye surgery in both eyes using the PRESBYOND method.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving binocular uncorrected near visual acuity (UNVA) of 0.1 logMAR or better | 6 months after surgery
  The primary endpoint of the study is the proportion of patients achieving a binocular uncorrected near visual acuity (UNVA) of 0.1 logMAR or better at 6 months postoperatively. Near visual acuity is assessed using standardized near vision charts under controlled lighting conditions, following standard clinical protocols. Measurements are taken binocularly to reflect functional vision in daily life.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - Eye Laser Specialists, Melbourne, VIC/Australia
  - Crystal Eye and laser Center, Craigie, Western Australia
- The Wellington Eye Centre, Wellington, New Zealand, New Zealand